CLINICAL TRIAL: NCT01312571
Title: Functional Magnetic Resonance Imaging (fMRI) and Treatment of Social Phobia Over the Internet: Cognitive Behavioural Therapy (CBT) Versus Computerized Attention Training and the Possible Effect of Genetic Variation. (SOFIE-8)
Brief Title: Treatment of Social Phobia Over the Internet
Acronym: SOFIE-8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Per Carlbring, PhD, Professor, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-185-31 M
Record Dates: First submitted 2010-08-31; First posted 2011-03-10 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Social Phobia
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive behavior therapy via the internet (Active Comparator): Cognitive behavior therapy via the internet with therapist support.
  Interventions: Behavioral: Internet-based cognitive behavioural therapy (iCBT)
- Attentional retraining (Active Comparator): Attentional retraining as described by Nader Amir.
  Interventions: Behavioral: Internet-based computerized attention training

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioural therapy (iCBT) — The Internet-based cognitive behavioural therapy (iCBT) consists of our structured self-help program lasting a total of nine active treatment weeks. This treatment program has been well evaluated and involved in several research projects.
  Arms: Cognitive behavior therapy via the internet
Behavioral: Internet-based computerized attention training — The Internet-based computerized attention training program lasting a total of four active treatment weeks. The treatment is consist of two training sessions per week, about 10 minutes long.
  Arms: Attentional retraining

SUMMARY:
Forty-eight people diagnosed with social phobia in an experimental study that randomized into two treatment groups: 1) Internet-based Cognitive Behavioural Therapy (iCBT) (n = 24) or 2) computerized attention training (n = 24). After nine weeks we change the condition of the two groups of research participants, which should therefore be given both treatments. Pre-and post measurement of functional magnetic resonance imaging (fMRI) will take place in the first round of treatment. Genotyping based on saliva samples takes place before the start of treatment, at the first fMRI measurement, for those who voluntarily leave the sample.

Study hypothesis

How is the brain activity of emotional processing and anxiety affected after completing an Internet-based CBT compared with computerized attention training? Does the treatment response of an Internet based treatment affects by variations in serotonin-transporter-linked promoter region (5-HTTLPR) and tryptophan hydroxylase-3 (TPH3) genes?

How is the genetic variations related to symptoms in social phobia (pre treatment)?

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet criteria for social phobia using the International classification system Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV).

Exclusion Criteria:

* Individuals with current depression and/or is suicide prone will be excluded from the study.
* With fMRI the following criteria must not be filled: previous surgery in the heart or brain, metals implanted in the body, dental braces or bridge; piercings that can´t be taken out, tattoos (shoulders, arms and back is not so good, the legs are okay if it is not too large); trouble to lie still for about an hour, pregnancy or history of neurological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Differences in recruited brain regions measured using regional cerebral blood flow | pretreatment (week 0), post treatment (week 11), 1 yr follow-up (week 63)
  Blood-oxygen-level dependence (BOLD) signal change as measured with 3.0 T fMRI
  Change from baseline in BOLD signal expected between time frames.
Social Phobia Screening Questionnaire (SPSQ) | pretreatment (week 0), post treatment (week 11), 1 yr follow-up (week 63)
  Social Phobia Screening Questionnaire (SPSQ), diagnostic tool for social phobia.
  Change from baseline in social anxiety symptoms expected between time frames.
Liebowitz Social Anxiety Scale self rated version (LSAS-SR) | pretreatment (week 0), post treatment (week 11), 1 yr follow-up (week 63)
  Measure social anxiety and social phobia.
  Change from baseline in social anxiety symptoms expected between time frames.
Social Interaction Anxiety Scale (SIAS) | pretreatment (week 0), post treatment (week 11), 1 yr follow-up (week 63)
  Measure social anxiety and social phobia.
  Change from baseline in social anxiety symptoms expected between time frames.
Social Phobia Scale (SPS) | pretreatment (week 0), post treatment (week 11), 1 yr follow-up (week 63)
  Measure social phobia.
  Change from baseline in social anxiety symptoms expected between time frames.

SECONDARY OUTCOMES:
Variation in genes that have been associated with emotional processing | pretreatment (week 0).
  We will study allelic variation in genes that have been associated with emotional processing e.g. monoaminergic gene polymorphisms such as the serotonin-transporter-linked promoter region (5-HTTLPR), tryptophan hydroxylase-2 (TPH2) G-703T, and Catechol-O-methyltransferase (COMT) 158Val/Met polymorphism
Montgomery Åsberg Depression Rating Scale (MADRS-S) | pretreatment (week 0), post treatment (week 11), 1 yr follow-up (week 63)
  Measure depression.
  Change from baseline in depressive symptoms expected between time frames.
Beck Anxiety Inventory (BAI) | pretreatment (week 0), post treatment (week 11), 1 yr follow-up (week 63)
  Measure anxiety.
  Change from baseline in anxiety symptoms expected between time frames.
Quality of Life Inventory (QOLI) | pretreatment (week 0), post treatment (week 11), 1 yr follow-up (week 63)
  Measure quality of life.
  Change from baseline in quality of life expected between time frames.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, Professor, Study Director — Umeå University; Gerhard Andersson, Professor, Study Chair — Linkoeping University; Tomas Furmark, Ass. professor, Study Chair — Uppsala University; Carl-Johan Olsson, Post doc, Study Chair — Umeå center for Functional Brain Imaging; Owe Bodlund, Ass. professor, Study Chair — NUS; Kristoffer NT Månsson, Student, Study Chair — Umeå University
Locations (1):
- Department of Psychology, Umeå University, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Background] Mansson KN, Frick A, Boraxbekk CJ, Marquand AF, Williams SC, Carlbring P, Andersson G, Furmark T. Predicting long-term outcome of Internet-delivered cognitive behavior therapy for social anxiety disorder using fMRI and support vector machine learning. Transl Psychiatry. 2015 Mar 17;5(3):e530. doi: 10.1038/tp.2015.22. PMID 25781229
- [Result] Mansson KN, Salami A, Frick A, Carlbring P, Andersson G, Furmark T, Boraxbekk CJ. Neuroplasticity in response to cognitive behavior therapy for social anxiety disorder. Transl Psychiatry. 2016 Feb 2;6(2):e727. doi: 10.1038/tp.2015.218. PMID 26836415
- [Result] Mansson KN, Carlbring P, Frick A, Engman J, Olsson CJ, Bodlund O, Furmark T, Andersson G. Altered neural correlates of affective processing after internet-delivered cognitive behavior therapy for social anxiety disorder. Psychiatry Res. 2013 Dec 30;214(3):229-37. doi: 10.1016/j.pscychresns.2013.08.012. Epub 2013 Sep 21. PMID 24064198